CLINICAL TRIAL: NCT07292688
Title: A Phase I, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of CM383 Following Intravenous and Subcutaneous Administration in Healthy Adult Subjects
Brief Title: Study of CM383 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM383-100002
Record Dates: First submitted 2025-12-03; First posted 2025-12-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CM383 subcutaneous injection group 1 (Experimental)
  Interventions: Biological: CM383
- CM383 subcutaneous injection group 2 (Experimental)
  Interventions: Biological: CM383
- CM383 intravenous infusion group (Experimental)
  Interventions: Biological: CM383

INTERVENTIONS:
Biological: CM383 — CM383 subcutaneous injection, once.
  Arms: CM383 subcutaneous injection group 1; CM383 subcutaneous injection group 2
Biological: CM383 — CM383 intravenous infusion, once.
  Arms: CM383 intravenous infusion group

SUMMARY:
This study is a Phase I, single-center, randomized, open-label, parallel-controlled study, aimed at evaluating the pharmacokinetics, pharmacodynamics, immunogenicity, safety, and tolerability of a single dose of CM383 administered via intravenous infusion or subcutaneous injection in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age ≥ 18 years & ≤54 years.
* Subjects voluntarily signed the Informed Consent Form and were able to comply with the provisions of this protocol.

Exclusion Criteria:

* The average number of cigarettes smoked per day is greater than 5 within 3 months prior to screening.
* Drinking heavily within 3 months prior to screening, or unable to guarantee not to drink alcohol during the research period, or positive alcohol breath testing.
* History of drug abuse within 1 year prior to screening, or positive urine drug abuse screening.
* Blood donation or any other form of blood loss exceeding 400 mL, or accepting blood transfusion within 12 weeks prior to screening.
* Suspected allergy to Aβ-antibody drugs, humanized monoclonal antibody drugs and their excipients, or other biological agents, or have a history of severe allergic reactions to other drugs.
* Severe trauma or undergo major surgery within 6 months prior to screening, or planned surgery during the research period.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic characteristics of a single-dose administration of CM383 in healthy male subjects | Up to Day 85
  Pharmacokinetic concentrations in serum and pharmacokinetic parameters: maximum concentration (Cmax).

CONTACTS AND LOCATIONS:
Overall Officials: Bo Jiang, Principal Investigator — The Second Affiliated Hospital Zhejiang University School of Medcine
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medcine, Hangzhou, China